CLINICAL TRIAL: NCT03975556
Title: Culturally-Adapted Diet for Puerto Rican Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: FDI Clinical Research (Other)
Responsible Party: Principal Investigator, Josiemer Mattei, Assistant Professor of Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB19-0184
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Hypertension; Dyslipidemias; High Triglycerides; High Blood Glucose; Abdominal Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Hypertension; Dyslipidemias; Hypertriglyceridemia; Hyperglycemia; Obesity, Abdominal | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be unaware of the which educational messages are considered intervention or control. Investigators will not be in contact with participants and will only receive coded data. Outcome assessor will be unaware of treatment allocation of participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group consisting of culturally-appropriate foods and diet advice in an initial individual session followed by daily text messages for 2 months (delivery phase). A reinforcement phase of 2-months will follow to repeat the text messages.
  Interventions: Behavioral: Culturally tailored food and diet advice
- Control (Active Comparator): Control arm of standard portion-control general nutritional and cooking advice at the initial individual session, followed by text messages for 2 months. A reinforcement phase of 2-months will follow to repeat the education and text messages.
  Interventions: Behavioral: Standard healthy eating advice

INTERVENTIONS:
Behavioral: Culturally tailored food and diet advice — Puerto Rico-tailored education includes strategies for healthy eating, preferences for traditional healthy foods, recommendations for limiting unhealthy traditional foods, portion sizes, etc.
  Arms: Intervention
Behavioral: Standard healthy eating advice — Standard healthy eating education includes strategies, foods, portions, and cooking and eating tips included in the My Plate dietary recommendations
  Arms: Control

SUMMARY:
This pilot project will determine whether a diet culturally-adapted to Puerto Ricans can effectively decrease cardiometabolic risk for diabetes. This will help define a culturally-appropriate, feasible, and sustainable diet intervention aimed at reducing type 2 diabetes and obesity outcomes.

DETAILED DESCRIPTION:
This pilot intervention will culturally-tailor a diet to the Puerto Rican adult population based on staple foods as well as culturally-appropriate strategies to reduce cardiometabolic risk factors of type 2 diabetes and obesity. Based on preliminary results from studies in the island, investigators will conduct a 4-month, 2-arm intervention among 200 adults (100 per arm) ages 25-65 living in Puerto Rico with at least 2 of 5 cardiometabolic risk factors. The two arms are: (1) intervention group consisting of culturally-appropriate advice in an initial individual session with daily text messages for 2 months (delivery phase); (2) control arm of standard general nutritional advice at the initial individual session, and text messages for 2 months. A reinforcement phase of 2-months will follow to repeat the education and text messages. Investigators will measure changes in cardiometabolic risk factors and in eating-behaviors and psychological measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-65 y old at the time of enrollment
2. Non-institutionalized
3. Living in PR at the time of recruitment and for at least the previous year and not planning to move from the island within the next 6 months
4. Able to answer questions without assistance
5. Having a cellphone with the capacity to receive text messages
6. Having at least two of the following:

   1. elevated BMI
   2. elevated waist circumference
   3. self-reported physician-diagnosed hypertension or use of hypertension medication or measured high blood pressure
   4. self-reported physician-diagnosed pre-diabetes or measured pre-diabetes
   5. self-reported physician-diagnosed dyslipidemia or use of lipid-lowering agents or laboratory values confirming dyslipidemia

Exclusion Criteria:

1. Under 25 or over 65 years of age
2. Currently do not live in Puerto Rico or have not lived in PR for at least 1 year or plan to move within 6 months
3. Institutionalized
4. Not able to answer questions without assistance
5. Not having at least 2 of the five listed metabolic criteria
6. Self-reported physician-diagnosed type 1 or type 2 diabetes or use of diabetes medication (including insulin), or diabetes-diagnosis values confirmed by laboratory.
7. Self-reported pregnancy
8. Gastrointestinal or chronic conditions
9. Food intolerance or allergies

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of dysregulated cradiometabolic risk factors | 4 months
  Estimate the change in the number of dysregulated cradiometabolic risk factors (outside of normal values)
Change in levels of adipose risk factor | 4 months
  Estimate the change in the value of waist circumference (cm)
Change in levels of blood pressure risk factors | 4 months
  Estimate the change in the value of systolic and diastolic blood pressure (mmHg)
Change in levels of metabolic risk factors | 4 months
  Estimate the change in the value of glucose, HDL, and triglycerides (mg/dL)

SECONDARY OUTCOMES:
Changes in diet quality score | 4 months
  Determine the change in score of short diet quality screener (range 18-54; from lowest to highest quality)
Changes in diet satisfaction: diet satisfaction scale | 4 months
  Determine the change in the score of the Diet Satisfaction Questionnaire (DSat-45) (range 45-225; from lowest to highest satisfaction) and its summed seven subscales (ranges 5-40)

CONTACTS AND LOCATIONS:
Overall Officials: Jose F Rodriguez Orengo, PhD, Study Director — FDI Clinical Research; Josiemer Mattei, PhD, MPH, Principal Investigator — Harvard Chan School of Public Health
Locations (1):
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
IPD will be managed and distributed observing NIH and IRB policies on the dissemination and sharing of research results. Study information and requests for data will be available immediately upon the data being de-identified and properly revised for quality control by contacting study investigators.
Supporting Information: Study Protocol, ICF
Time Frame: 1-year
Access Criteria: The requested data will be shared with investigators via a secured, password-protected software website, upon request.

REFERENCES:
- [Derived] Mattei J, Diaz-Alvarez CB, Alfonso C, O'Neill HJ, Rios-Bedoya CF, Malik VS, Godoy-Vitorino F, Cheng C, Spiegelman D, Willett WC, Hu FB, Rodriguez-Orengo JF. Design and Implementation of a Culturally-Tailored Randomized Pilot Trial: Puerto Rican Optimized Mediterranean-Like Diet. Curr Dev Nutr. 2022 Dec 23;7(1):100022. doi: 10.1016/j.cdnut.2022.100022. eCollection 2023 Jan. PMID 37181130